CLINICAL TRIAL: NCT06454097
Title: Study on Radiogenomics Features Associated With Radiochemotherapy Sensitivity in Gliomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 82072786
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluate the response of patients with glioma to radiochemotherapy (Other): The response of patients with glioma to radiochemotherapy will be assessed by the RANO criteria and the established radiogenomics-based artificial intellegent model.
  Interventions: Diagnostic Test: Assess the response glioma to radiochemotherapy using radiogenomics-based AI model

INTERVENTIONS:
Diagnostic Test: Assess the response glioma to radiochemotherapy using radiogenomics-based AI model — Predict the radiochemotherapy sensitivity of patients with glioma using an established radiogenomics-based artificial intellegent mode

SUMMARY:
The MRI data were collected from patients with gliomas before surgery, 2 weeks before initiating radiochemotherapy, 1 month after completing the radiotherapy (for lower-grade gliomas, LGG), or 4 and 10 months after completing the radiochemotherapy (for high-grade gliomas, HGG). Radiochemotherapy sensitivity labels were constructed based on the MRI images obtained before and after radiochemotherapy, following the RANO criteria. Radiomics features were extracted from preoperative MRI images and combined with transcriptomic information obtained from tumor tissue sequencing. This process allowed the construction of a radiogenomics model capable of predicting the response of gliomas to radiochemotherapy.

In this prospective cohort study, we will recruit patients with gliomas who have undergone craniotomy and received postoperative radiotherapy or radiochemotherapy (in cases of LGG and HGG, respectively). MRI images of the same sequences will be collected at corresponding time points, and transcriptomic sequencing will be performed on tumor tissue obtained during surgery. The established model will be applied to predict radiochemotherapy sensitivity and compared with the 'true' radiochemotherapy sensitivity labels, which are constructed based on the RANO criteria, to evaluate the predictive performance of the model.

DETAILED DESCRIPTION:
This trial aims to recruit 100 cases of LGG and 100 cases of HGG based on statistical calculations. MRI data, including T1-weighted, T2-weighted, T1 contrast-enhanced, and T2-Fluid Attenuated Inversion Recovery (FLAIR) sequences, will be collected before surgery, 2 weeks before initiating radiochemotherapy, 1 month after completing the radiotherapy (LGG), or 4 and 10 months after completing the radiochemotherapy (HGG).

The collected MRI images before and after radiochemotherapy will be used to assess changes in tumor volume. The RANO criteria will be employed to determine the tumor's sensitivity to radiochemotherapy: a complete response and partial response will be classified as sensitive, while stable disease and disease progression will be considered insensitive.

Radiomics features will be extracted using the open-source 'PyRadiomics' python package after performing image preprocessing and segmentation. Transcriptomic data will be obtained by conducting RNA sequencing analysis on tumor samples collected during surgery. Selected radiogenomic features will be incorporated into a pre-constructed machine learning model to predict the sensitivity of gliomas to radiochemotherapy. The model's performance will be evaluated using metrics such as classification accuracy (ACC), area under the receiver operating characteristic curve (AUC), positive predictive value (PPV), and negative predictive value (NPV).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Histologically confirmed glioma
* No history of other brain tumors or previous cranial surgeries
* No history of preoperative radiotherapy or chemotherapy
* Available preoperative, pre-radiotherapy(postoperatively), and post-radiotherapy magnetic resonance imaging (MRI) data

Exclusion Criteria:

* Those who do not meet any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the AI model in predicting radiochemotherapy respone | 1 month after radiotherapy (LGG); 4 and 10 months after radiochemotherapy (HGG)
  Sensitivity = TP/(TP+FN)
Specificity of the AI model in predicting radiochemotherapy respone | 1 month after radiotherapy (LGG); 4 and 10 months after radiochemotherapy (HGG)
  Specificity = TN/(TN+FP)
Area under the Receiver Operating Characteristic curve (AUC) | 1 month after radiotherapy (LGG); 4 and 10 months after radiochemotherapy (HGG)
  AUC measures the entire two-dimensional area underneath the entire ROC curve

SECONDARY OUTCOMES:
Accuracy of the AI model in predicting radiochemotherapy respone | 1 month after radiotherapy (LGG); 4 and 10 months after radiochemotherapy (HGG)
  Accuracy of radiotherapy sensitivity prediction AI model = (TP+TN)/ (TP+TN +FP+FN)
Positive predictive value (PPV) of the AI model in predicting radiochemotherapy respone | 1 month after radiotherapy (LGG); 4 and 10 months after radiochemotherapy (HGG)
  PPV of radiotherapy sensitivity prediction AI model = [TP/(TP+FP)]*100
Negative predictive value (NPV) of the AI model in predicting radiochemotherapy respone | 1 month after radiotherapy (LGG); 4 and 10 months after radiochemotherapy (HGG)
  NPV of radiotherapy sensitivity prediction AI model = [TN/(FN+TN)]*100

CONTACTS AND LOCATIONS:
Overall Officials: Yinyan Wang, MD and PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China